CLINICAL TRIAL: NCT02423525
Title: A Phase I Dose Escalation and Central Nervous System (CNS) Pharmacokinetic Study of the ErbB Family Inhibitor Afatinib in Patients With Recurrent or Progressive Brain Cancer
Brief Title: Safety Study of Afatinib for Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santosh Kesari (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Santosh Kesari, Director, Neuro-Oncology, Saint John's Cancer Institute
Organization: Saint John's Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.229; 20161975 (Other: Western Institutional Review Board)
Record Dates: First submitted 2015-02-05; First posted 2015-04-22 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Brain Cancer
Keywords: glioblastoma; astrocytoma; oligodendroglioma; mixed oligoastrocytoma; low grade gliomas; brain metastases; meningiomas; leptomeningeal metastases
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Meningioma; Meningeal Carcinomatosis | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afatinib (Experimental): Afatinib tablets are taken by mouth. Dose Level 1: 80 mg every 4 days Dose Level 2: 120 mg every 4 days Dose Level 3: 180 mg every 4 days Dose Level 4: 280 mg every 7 days
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib
  Other Names: Gilotrif

SUMMARY:
The purpose of this study is to try to determine the maximum safe dose of afatinib that can be administered to people with brain cancer. Other purposes of this study are to:

* find out what effects (good and bad) afatinib has;
* see how much drug gets into the body by collecting blood and cerebrospinal fluid for use in pharmacokinetic (PK) studies;
* learn more about how afatinib might affect the growth of cancer cells;
* look at biomarkers (biochemical features that can be used to measure the progress of disease or the effects of a drug).

DETAILED DESCRIPTION:
This is an open-label, single institution, Phase I 3+3 dose escalation study to describe the safety and tolerability of afatinib in patients with brain cancer having failed prior therapy and to determine the recommended phase II dose.

Eligible patients will receive afatinib in treatment cycles of 28 days that will consist of afatinib administered orally by mouth once every four days. Patients will be assigned to the dose level open at the time of their enrollment. Patients will continue dosing of afatinib until disease progression, unacceptable toxicity, withdrawal of consent, or treating physician determines it is in their best interest to stop. Guidelines for modifying study drug doses is provided for the management of adverse treatment effects.

All patients will have regular evaluations for assessment of safety parameters as detailed in the study flow chart. Lumbar puncture and blood draw for assessing afatinib levels will occur as detailed in the study flow chart.

Neurological imaging and assessment for response will be performed approximately every eight weeks. Tumor response will be assessed according to Response Assessment in Neuro-Oncology (RANO) Working Group criteria.

An end of treatment evaluation will occur when a patient permanently discontinues study drug, as detailed in the study flow chart. Patients will then be followed every four months for survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis

  1. Dose Escalation Cohorts: Histologically confirmed diagnosis of brain cancer:

     1. glioblastoma (GBM),
     2. anaplastic astrocytoma (AA),
     3. anaplastic oligodendroglioma (AO),
     4. anaplastic mixed oligoastrocytoma (AMO),
     5. low grade gliomas,
     6. brain metastases,
     7. meningiomas,
     8. leptomeningeal metastases
     9. chordomas
     10. pituitary tumors
     11. medulloblastomas
  2. Expansion Cohort: Histologically confirmed diagnosis of high-grade glioma with altered EGFR (e.g., amplification, mutation), including:

     1. glioblastoma (GBM),
     2. anaplastic astrocytoma (AA),
     3. anaplastic oligodendroglioma (AO),
     4. anaplastic mixed oligoastrocytoma (AMO)
* Has failed prior standard therapy including maximal safe surgical resection (when appropriate for the specific cancer type), radiation therapy (when appropriate for the specific cancer type), and systemic therapy (when appropriate for the specific cancer type).
* For diagnosis of GBM: has undergone maximal safe surgical resection, a course of postoperative radiation therapy with concurrent temozolomide, and maintenance temozolomide.
* For diagnosis of meningioma: has no other option of standard therapy such as surgical resection (partial or total resection) or radiation.
* Age 18 years and older.
* Karnofsky Performance Status ≥ 60%.
* Adequate organ function, defined as all of the following:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  2. Platelet count ≥ 100 x 109/L.
  3. Hemoglobin ≥ 9.0 g/dL.
  4. Total Bilirubin ≤ 1.5 institution's upper limit of normal (ULN).
  5. Aspartate amino transferase (AST) ≤ 2.5 x institution's ULN.
  6. Alanine amino transferase (ALT) ≤ 2.5 x institution's ULN.
  7. Alkaline phosphatase (ALP) ≤ 2.5 x ULN unless considered tumor related.
* Recovered from any previous therapy-related toxicity to Grade 1 or to their clinical baseline at study entry.
* Women of child-bearing potential has negative serum or urine pregnancy test before the initiation of study drug dosing.

Exclusion Criteria:

* Insufficient time from prior therapy to study entry:

  1. less than 28 days from whole-brain radiotherapy (WBRT) or stereotactic radiosurgery (SRS);
  2. less than 28 days from any investigational agent;
  3. less than 28 days from prior cytotoxic therapy (except 23 days from prior temozolomide, 14 days from vincristine (for GBM: 14 days from irinotecan or topotecan), 42 days from nitrosoureas, 21 days from procarbazine, irinotecan or topotecan administration);
  4. less than 14 days from hormonal treatment
  5. less than 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc.
  6. When radiation necrosis is suspected, standard of care confirmatory imaging, such as MRI perfusion, magnetic resonance (MR) spectroscopy and or PET will be performed, and patients with findings consistent with radiation necrosis will be excluded.
* Current or anticipated use of enzyme-inducing anti-epileptic drugs (EIAED).
* Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study.
* Known hypersensitivity to afatinib or its excipients.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3 or 4, unstable angina or poorly controlled arrhythmia, or myocardial infarction within 6 months prior to enrollment.
* Pregnant, nursing, or not using acceptable method of birth control.
* Any history of or concomitant condition that would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug.
* Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
* Known pre-existing interstitial lung disease.
* Known active hepatitis B infection (defined as presence of Hep B sAg and/ or Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.
* Prior participation in a blinded afatinib clinical study, even if not assigned to afatinib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities of pulsatile afatinib | first 28 days of treatment
  Number of side effects of study treatment that prevent an increase in dose or level of that treatment
Maximum tolerated dose (MTD) of pulsatile afatinib | first 28 days of treatment
  The highest dose evaluated that does not cause unacceptable side effects

SECONDARY OUTCOMES:
Treatment-emergent adverse events | 7 months
  Type, number, grade and seriousness of adverse events reported after the first dose of study treatment
Afatinib levels in cerebrospinal fluid (CSF) and blood | 52 days
  Measurement of afatinib concentration in CSF and blood at defined timepoints
Objective response rate as assessed by the RANO criteria | approximately 6 months to 1 year
  Tumor response compared to baseline as assessed by the RANO criteria
Best overall response rate | approximately 6 months to 1 year
  Best tumor response compared to baseline
Progression free survival | up to 5 years
  Time between the start of treatment to disease progression
Overall Survival | up to 5 years
  Time between the start of treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided